CLINICAL TRIAL: NCT00832364
Title: Randomized, Controlled Trial of an Injectable Biologic and U0279 as Combination Therapy for Severe Plaque-Type Psoriasis
Brief Title: Trial of an Injectable Biologic and U0279 as Combination Therapy for Severe Plaque-Type Psoriasis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Business decision. No patients were enrolled
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114549; U0279-401
Record Dates: First submitted 2009-01-27; First posted 2009-01-30 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2011-06

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis; Moderate to Severe Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Acitretin; Etanercept

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): U0279 and Injectable Biologic
  Interventions: Drug: Acitretin (also called U0279); Biological: Etanercept
- 2 (Placebo Comparator): Placebo and Injectable Biologic
  Interventions: Drug: Placebo; Biological: Etanercept

INTERVENTIONS:
Drug: Acitretin (also called U0279) — Capsules containing 25 mg U0279 taken once a day.
  Arms: 1
Drug: Placebo — Placebo capsules
  Arms: 2
Biological: Etanercept — Injectable Biologic
  Other Names: Embrel

SUMMARY:
The purpose of the study is to assess the safety and efficacy of an injectable biologic and U0279 as combination therapy compared to that of an injectable biologic alone for severe plaque-type psoriasis.

DETAILED DESCRIPTION:
The study is being conducted in order to obtain safety and efficacy data for an injectable biologic and U0279 as combination therapy compared to that of an injectable biologic alone for severe plaque-type psoriasis. The subjects will be randomized to either U0279 or placebo after having been on an injectable biologic for 12 weeks previously. The subject will be on study medication for 12 weeks. The subjects must have moderate to severe Psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 18 years of age or older.
* Surgically sterile females. Females who have had a hysterectomy or completed menopause are allowed.
* Affected Body Surface Area with psoriasis of ≥10%.
* Psoriasis Global Assessment rating of "moderate to severe" or "severe".
* Achieved mild to moderate improvement after receiving an injectable biologic therapy for at least 12 weeks.
* A PASI score of ≥ 50 and ≤75
* Capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol specific procedures are performed

Exclusion Criteria:

* Understand that the sponsor can not pay for the an injectable biologic therapy during the course of the study; be willing to pay out of pocket or secure payment through their private health insurance for an injectable biologic.
* History of systemic infection, or other conditions that may interfere with study evaluations or may increase risk for participation. such as, tuberculosis, human immunodeficiency virus (HIV), hepatitis; congestive heart failure or demyelinating disorder.
* Used of prohibited medications or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Primary endpoints - Mean change in % BSA psoriasis involvement from baseline to week 12 and the mean change in PASI score from baseline to Week 12. | Baseline & Week 12

SECONDARY OUTCOMES:
Mean change from baseline in PGA at week 12, % of subjects with improvement in PASI 50 to 75 from baseline to week 12 and % of subjects with improvement in PASI 75 to 90 from baseline to week 12. | Baseline & Week 12

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - UCSF - Dermatology Psoriasis & Skin Treatment Center, San Francisco, California
  - Physicians Skin Care, Louisville, Kentucky
  - Mt. Sinai School of Medicine Department of Dermatology, New York, New York